CLINICAL TRIAL: NCT02844842
Title: Evaluation of Tolerability and Safety of "Allergovac Poliplus" in Polysensitized Patients With Rhinitis or Allergic Rhinoconjunctivitis With or Without Asthma: A Study in Daily Clinical Practice
Acronym: APOLO
Status: Completed | Type: Observational
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: BIA-ALE-2016-01
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Allergic Rhinitis; Rhinoconjunctivitis; Asthma
Keywords: mild or moderate
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 day initiation schedule: The initiation Schedule consists in administering 0.2 mL and 0.3 mL with 30 minutes of interval in the same day. Thus, the patient will reach the maintenance dose of 0.5 mL in one day.
  Interventions: Biological: Allergovac Poliplus
- Rapid initiation schedule: The patient will receive 3 increasing doses (0.1 mL + 0.3mL + 0.5 mL) weekly doses till the maintenance dose (0.5 mL) is reached.
  Interventions: Biological: Allergovac Poliplus

INTERVENTIONS:
Biological: Allergovac Poliplus

SUMMARY:
This is an observational prospective study to assess the tolerability and safety of treatment of SCIT Allergovac Poliplus polymerized in depot presentation. The study drug will be administered either by a 1 day Schedule or by a rapid Schedule (3 increasing weekly doses at initiation period till maintenance dose is reached) The study population is both: adult and child, polysensitized to at least 2 allergen sources with rhinitis or allergic rhinoconjunctivitis. Patients may also present a concomitant mild or moderate asthma.

The assignment of a patient to a particular therapeutic strategy will not be decided in advanced by a trial protocol but will be determined by routine clinical practice. The decision of the investigator to prescribe a particular treatment will be clearly dissociated from the decision to include the patient in the study. The patients will not suffer any intervention, whether diagnostic or monitoring, other than the usual in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 5 and 60 years who present rhinitis or allergic rhinoconjunctivitis caused by IgE-mediated sensitization to more than one allergen source with or without mild / moderate asthma.
2. Patients eligible for immunotherapy treatment with Allergovac Poliplus according to investigator criteria.
3. Patients must provide written informed consent. It is the case of children , the legal representative or tutor of the child must sign the inform consent form.

Exclusion Criteria:

1. Patients that according to the investigator criteria may present difficulties for understanding the patient information sheet, completing the questionnaires and self-administered scales.
2. Patients that according to the investigator may present difficulties to complete the patient diary.
3. Patients who are participating in another clinical trial or observational study.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Polisensitized patients with allergic rinitis and rhinoconjunctivitis with or without associated mild or moderate asthma
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2016-11-23; Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse drug reactions | From patient ICF signature till 1 week after last administered dose

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - C.H.U A Coruña, A Coruña
  - Hopsital de Vinalopó, Elche
  - Clínica Dr. Arias Irigoyen, Huelva
  - Clínica Dra. Victoria Moreno, Huelva
  - Hospital de Lugo, Lugo
  - Clínica de Asma y Alergia Dres. Ojeda, Madrid
  - Hospital Principe de Asturias, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital de Onteniente, Ontinyent
  - Hospital de Tórax, Santa Cruz de Tenerife
  - Hospital Ntra. Sra de la Candelaria, Santa Cruz de Tenerife
  - Hospital Joan XXIII, Tarragona
  - Hospital de Terrassa, Terrassa
  - Hospital de Manises, Valencia
  - Hospital de Xátiva, Xátiva